CLINICAL TRIAL: NCT05779813
Title: Genetic Frontotemporal Dementia Initiative for Neurodevelopment
Acronym: GENFI-NeuroDev
Status: Recruiting | Type: Observational
Sponsor: Western University (Other)
Responsible Party: Principal Investigator, Dr. Elizabeth Finger, Director of Research, Dept. of Clinical Neurological Sciences, Western University
Other Study IDs: GENFI-NeuroDev
Record Dates: First submitted 2023-02-27; First posted 2023-03-22 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Frontotemporal Dementia; Family Members
MeSH Terms: conditions — Frontotemporal Dementia

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is an international multi-centre cohort study of first and second degree family members of individuals who carry Frontotemporal Dementia (FTD) mutations in MAPT, GRN or C9ORF72 repeat expansions for youths between the ages 9-17.

DETAILED DESCRIPTION:
GENFI-NeuroDev will study genetic FTD and its associated disorders (including Motor Neurone Disease (MND)/Amyotrophic Lateral Sclerosis(ALS)) in members of families with a known mutation in GRN or MAPT or an expansion in C9orf72. Participants with at-risk members of families (first-degree and second-degree relatives of known genetic mutation carriers). All GENFI-NeuroDev participants will be assessed longitudinally with a set of clinical, neuropsychiatric, cognitive, imaging and biosample protocols. Parents or guardians of potential GENFI NeuroDev participants are all aware of the autosomal dominant genetic nature of FTD in their family prior to being approached for potential participation in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained and documented (from the participant and their substitute decision maker). This can be obtained in person or remotely.
2. Youths between the ages of 9 and 16 inclusive at time of enrollment, followed until age 17.
3. Youths must have a 1st or 2nd degree biological relative who has participated (past or present) in the Genetic Frontotemporal Dementia Initiative (GENFI) study or with genetic FTD (i.e. a known mutation in biological parent or grandparent).
4. Parent(s)/guardian deem appropriate to participate.
5. Must have a study partner who can participate as required in the protocol (provide corroborative information). Study partner must have regular contact with the participant and must be parent/guardian of this participant.
6. Must have age-appropriate awareness that FTD runs in their family as determined by local PI.

Exclusion Criteria:

1. Current structural brain abnormality affecting cognition or behaviour not thought to be possibly related to genetic FTD that would prevent completion of study assessments (such as brain tumor, stroke, hydrocephalus).
2. Other concerns that participation in the study may not be in the best interest of the youth or parent, as raised by the participant's parent/guardian/primary care provider, local site PI or psychologist.
3. Lack of study partner.
4. For MRI: meeting any MRI incompatible criteria. Note: Participants may opt to decline MRI scans and complete the other measures.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Youths between the ages of 9 and 16 inclusive at time of enrollment who have a 1st or 2nd degree biological relative with genetic FTD (i.e. a known mutation in biological parent or grandparent). Parents or guardians of potential GENFI NeuroDev participants are all aware of the autosomal dominant genetic nature of FTD in their family prior to being approached for potential participation in this study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-03-31 (Actual); Primary Completion 2033-03 (Estimated); Study Completion 2035-03 (Estimated)

PRIMARY OUTCOMES:
Brain development as measured by structural and functional Magnetic Resonance Imaging | Through study completion, an average of 2 years

OTHER OUTCOMES:
Fluid biomarkers of neurodevelopment, neurodegeneration and inflammation | Through study completion, an average of 2 years
  To examine differences compared to age matched non-carriers in physiologic signals in fluid biomarkers of synaptic markers, axonal markers, and neuroinflammation markers.
Resting State quantitative electroencephalogram (EEG) | Through study completion, an average of 2 years
  To analyze resting state quantitative EEG (qEEG) power spectral density, a reliable metric of CNS physiology in children.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Finger, MD, Principal Investigator — Western University
Locations (1):
- Western University, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Data will be shared within the GENFI consortium based on specific data access requests.